CLINICAL TRIAL: NCT05060328
Title: Use of Google Translate to Enhance Patient Pain and Nausea Assessment and Satisfaction After General Anesthesia: A Pilot Feasibility Study
Brief Title: Use of Google Translate to Enhance Patient Pain and Nausea Assessment and Satisfaction After General Anesthesia
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-1345; NCI-2021-09116 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1345 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-09-15; First posted 2021-09-29 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Health services research (Google Translate Conversation Mode): Patients use Google Translate "Conversation Mode" translation application before and after surgery. Patients also complete survey over 10 minutes.
  Interventions: Other: Medical Device Usage and Evaluation; Other: Survey Administration

INTERVENTIONS:
Other: Medical Device Usage and Evaluation — Use Google Translate "Conversation Mode" translation application.
Other: Survey Administration — Complete survey

SUMMARY:
This study investigates the use of Google Translate "Conversation Mode" translation service to improve communication about pain and nausea with Spanish-speaking patients who are recovering after surgery. The Google Translate "Conversation Mode" translation application is designed to provide translation from one language to another and used to allow the nurse or study doctor to communicate with patients in Spanish by asking pre-prepared questions through an electronic device such as an iPad or iPhone. Google Translate "Conversation Mode" may facilitate assessment of pain and nausea after surgery in Spanish speaking patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the feasibility of Google Translate "Conversation Mode" use to assess postoperative surgical pain presence, location and intensity, and nausea presence and intensity in Spanish speaking patients in the post-anesthesia care unit (PACU).

SECONDARY OBJECTIVES:

I. To evaluate the length of stay in PACU. II. To assess patient satisfaction with regards to pain/nausea experienced in PACU.

III. To determine nursing satisfaction with regards to the use of Google Translate "Conversation Mode".

OUTLINE:

Patients use Google Translate "Conversation Mode" translation application before and after surgery. Patients also complete survey over 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Patients between 18-80 years of age whose primary language is Spanish and will require translation services as part of standard care
* American Society of Anesthesiologists physical status (ASA) 1-3
* Are scheduled surgery under general anesthesia
* Ability to understand and complete all study questionnaires

Exclusion Criteria:

* Emergency surgery
* ASA >= 4
* Patients who do not require official translation services for consent purposes
* Patients who have chronic pain and/or are taking opioids chronically (daily intake for more than a month before surgery)
* Patients who undergo craniotomy
* Patients with a hearing impairment that prevents the ability to hear the recorded statements; and/or a cognitive impairment that would prevent them from completing post-op assessments

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with scheduled surgery under general anesthesia and will require translation services as part of standard care
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Ability to respond to the questions when asked using Google Translate | 1 year
  The feasibility rate and its 95% confidence interval will be estimated.

CONTACTS AND LOCATIONS:
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org